CLINICAL TRIAL: NCT01437644
Title: Post-operative Pain in Children With Cerebral Palsy Following Major Hip Surgery: a Double Blind Randomised Placebo Controlled Trial of Pre-operative Botulinum Toxin Type A
Brief Title: The Post-Operative Pain in Cerebral Palsy (POPPIES) Trial
Acronym: POPPIES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Fabian Norman-Taylor, Consultant Orthopaedic Surgeon, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-023240-33; PB-PG-1208-18132 (Other Grant/Funding Number: NIHR RfPB grant (UK)); 2010-023240-33 (EudraCT Number); 11/WA/0010 (Other: Research Ethics Committee for Wales)
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Cerebral Palsy; Post-operative Pain
Keywords: Cerebral Palsy; Hip displacement; Hip surgery; Post-operative pain; Botulinum Toxin
MeSH Terms: conditions — Cerebral Palsy; Pain, Postoperative; Hip Dislocation | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum Toxin TypeA (Active Comparator): A single dose of active drug or placebo will be administered immediately prior to surgery.
  The injections will be given to the anaesthetised child before the surgical procedure begins. The surgeon will perform the injections at three muscle groups around each hip: the adductors, hamstrings and iliopsoas muscles. Two units per kilogram will be given at each site. The maximum dose will be 12 units per kilogram or 500 units in total (whichever is the lesser), divided equally between six or three sites. A total of 2 ml of isotonic saline will be used to dissolve the contents of the trial vial of Botox. Each active drug vial will contain 100 iu of the Botox preparation. The volume injected will be dependent on the weight of the child. Injections of normal saline will be administered in those children randomised to the placebo arm of the study.
  Interventions: Drug: botulinum toxin intramuscular injection
- Saline (Placebo Comparator): The injections will be given to the anaesthetised child before the surgical procedure begins. The surgeon will perform the injections at three muscle groups around each hip: the adductors, hamstrings and iliopsoas muscles. Injections of normal saline will be administered in those children randomised to the placebo arm of the study. The volume of normal saline injected will be equal to the volume of normal saline that would have been used if the child had been randomised to botulinum toxin. The injector will be blinded, as the solution is drawn up by unblinded nurses.
  Interventions: Drug: botulinum toxin intramuscular injection

INTERVENTIONS:
Drug: botulinum toxin intramuscular injection — A single dose of active drug or placebo will be administered immediately prior to surgery.
  The injections will be given to the anaesthetised child before the surgical procedure begins. The surgeon will perform the injections at three muscle groups around each hip: the adductors, hamstrings and iliopsoas muscles. Two units per kilogram will be given at each site. The maximum dose will be 12 units per kilogram or 500 units in total (whichever is the lesser), divided equally between six or three sites. Each active drug vial will contain 100 iu of the Botox preparation. The volume injected will be dependent on the weight of the child. Injections of normal saline will be administered in those children randomised to the placebo.
  Other Names: Botox, Allergan.

SUMMARY:
Cerebral palsy is common. It affects approximately 3 per 1000 children. Hip displacement due to muscle tightness (spasticity) occurs in up to half of the more severely affected children, and many of these children require major (bony) hip surgery. After bony hip surgery the management of pain is very difficult, as spasticity tends to increase and causes painful spasms which are difficult to control. Botulinum Toxin injections are known to reduce spasticity and therefore should also reduce pain. These injections take at least a week to work, but the effects can last for months. Botulinum Toxin is already an established treatment for chronic hip pain prior to surgery. The investigators aim to find out whether Botulinum Toxin injections can reduce post-operative pain. The identification of the level of pain can be challenging because most of these children are unable to communicate verbally. The investigators are therefore using a validated pain scoring tool that was designed especially for such children. This study will be the first to describe fully the pain experience of children with cerebral palsy undergoing this type of major surgery. The investigators will compare Botulinum Toxin injections with placebo (non-active) injections. There is a high emotional and financial burden on the families of these children. Families describe high levels of emotional distress around the time of surgery, particularly when their child is in pain. Difficulty with pain control post operatively may delay discharge from hospital and parental return to work. It causes disrupted sleep for the child and family and may delay the child's return to school. The results of this study will be shared with professionals and families at international conferences and in scientific and popular (patient-based) publications. This study cannot be undertaken in adults with cerebral palsy as they only rarely undergo this sort of surgery.

DETAILED DESCRIPTION:
Botulinum toxin injected intramuscularly is beneficial in the management of spasticity and as a treatment for chronic hip pain in children with cerebral palsy. Botulinum injections also seem to be useful in reducing spasticity in the acute post operative period; the benefits of botulinum toxin have been described in one study for post-operative pain following minor hip surgery. After major (bony) hip surgery these children experience significantly more pain, which also seems to be exacerbated by spasticity. Botulinum toxin may therefore reduce pain following major hip surgery. Research is required to assess its value in this setting. This cannot be studied in adults as they rarely undergo such surgery.

Cerebral palsy (CP) is the commonest cause of physical disability in childhood, it affects up to 3 children per 1000 throughout Europe (1;2). The Gross Motor Function Classification System (GMFCS) was designed for children and describes their level of motor skill (3). Over 25% of children with CP probably fall in the more severely affected groups - GMFCS levels IV and V. These children are not independently ambulant and are more likely to have cognitive and communication difficulties. They are at high risk of developing hip displacement (ie the hip gradually comes out of its socket) (4-10). Previous studies suggest that up to half of these hips are painful and it is well-established that hip displacement is painful for some children (14-18). Prevention of painful hip displacement has been advocated through screening programmes and timely surgical intervention (11-13). Some children need bony reconstructive surgery. Long term follow up studies have demonstrated that this maintains the position of the femoral head in the acetabulum over time, reducing the likelihood of a painful hip due to dislocation (9;10).

The management of pain in the severely neurologically impaired child undergoing hip (or any other) surgery is challenging and various strategies have been employed, including the use of post-operative epidurals. In a child with spasticity abnormally high post-operative muscle tone may be a cause painful muscle spasms. These involuntary and sustained muscle contractions are thought to contribute significantly to pain in children with cerebral palsy and a hip problem. There are a number of treatments available for muscle spasm in cerebral palsy; all are systemic except botulinum toxin which targets individual muscles by means of intramuscular injection. Botulinum toxin type A (BTXA) injection is a well established, clinically effective and safe treatment for muscle spasticity in CP (2;19;20). Research suggests it may have a beneficial effect in reducing pain due to spasticity (18). Graham and co-workers established that BTXA was safe in the perioperative period for children with cerebral palsy undergoing soft tissue surgery for a hip problem. Lundy and Fairhurst demonstrated BTXA is safe and effective in children with severe cerebral palsy, GMFCS IV&V when doses are given in line with the European Consensus guidelines. (24) Work on pain in children with CP suggests that anxiety and unrelieved pain may stimulate the autonomic nervous system in such a way that these children may actually have an amplified pain response when undergoing surgical procedures. Actions such as stretching muscles in a cast or for rehabilitation exercises may exacerbate spasms and therefore increase pain (8;17;21).

Describing pain in children with cognitive impairment however is challenging. Studies have focused on the report of pain symptoms, duration, intensity and analgesia requirements. Hunt et al provided a validated pain profile questionnaire which objectively measures pain in the more severely neurologically affected group of children with communication difficulties (22). The investigators have gained experience using this Paediatric Pain Profile to describe levels of pain in this group of children. It is a validated and user friendly system, already in place at this institution.

ELIGIBILITY:
Inclusion Criteria:

1. The child has displaced hips requiring bony orthopaedic surgery (osteotomy) due to cerebral palsy (appendix 2).
2. The child is between the ages of 2 and 15 years (inclusive).
3. The child has a GMFCS level of IV or V
4. The child has a diagnosis of hypertonic cerebral palsy (or a diagnosis consistent with this nomenclature)
5. The child does not communicate verbally
6. Informed consent to participate has been given by parent/carer.

Exclusion Criteria:

1. The child is younger than 2 years or older than 15 years
2. The child has an acute and current systemic infection or illness
3. The child has had botulinum toxin injections within the past 4 months
4. The child has had a previous reaction to botulinum toxin
5. The child has received or is likely to receive, at the time of trial drug or placebo administration, medications which might interact with botulinum toxin (this does not apply to any drugs at present)
6. Insufficient understanding of the trial by the parent or carer, in the investigator's opinion.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Paediatric Pain Profile | 6 weeks post-op
  The primary endpoint is the change in pain score during the six weeks following the operation. Pain will be measured using a validated questionnaire, the Paediatric Pain Profile. This scores pain by rating twenty different items of observed behaviour on an ordinal scale of 0 to 3 with a composite score of 0 to 60. It has been validated in children with severe cerebral palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Newton, Study Director — King's Health Partners Clinical Trials Office
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, London, United Kingdom